CLINICAL TRIAL: NCT00647530
Title: FOxTROT - Fluoropyrimidine, Oxaliplatin and Targeted Receptor Pre-Operative Therapy: a Controlled Trial in High-Risk Operable Colon Cancer
Brief Title: Fluorouracil and Oxaliplatin With or Without Panitumumab In Treating Patients With High-Risk Colon Cancer That Can Be Removed by Surgery
Acronym: FOxTROT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCTU-FOXTROT-001; CDR0000590089 (Registry Identifier: PDQ (Physician Data Query)); ISCRTN 87163246; EUDRACT 2007-001987-55; EU-20830; MREC-07/S0703/57; UKCRN 3771
Record Dates: First submitted 2008-03-28; First posted 2008-03-31 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage I colon cancer; stage II colon cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Panitumumab; Capecitabine; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Pre- plus Post-operative chemotherapy (+/- Panitumumab) vs standard post-operative chemotherapy.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pre&Post Op Chemo (Experimental): 12 weeks of OxFP neuoadjuvantly followed by surgery and 18 weeks of OxFP
  Interventions: Drug: capecitabine; Drug: fluorouracil; Drug: oxaliplatin
- Pre&Post Op Chemo with P-mab (Experimental): 12 weeks of OxFP and panitumumab neuoadjuvantly followed by surgery and 18 weeks of OxFP alone.
  Interventions: Biological: panitumumab; Drug: fluorouracil; Drug: oxaliplatin
- Post Op Chemo (Active Comparator): surgery followed by 24 weeks of OxFP.
  Interventions: Drug: capecitabine; Drug: fluorouracil; Drug: oxaliplatin

INTERVENTIONS:
Biological: panitumumab
  Arms: Pre&Post Op Chemo with P-mab
Drug: capecitabine
  Arms: Post Op Chemo; Pre&Post Op Chemo
Drug: fluorouracil
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether chemotherapy is more effective with or without panitumumab in treating patients with colon cancer.

PURPOSE: This randomized phase III trial assessing whether preoperative chemotherapy and/or an anti-EGFR monoclonal antibody improve outcome in high risk operable colon cancer.

DETAILED DESCRIPTION:
FOxTROT is a multi-centre randomised controlled trial (RCT) with the following objectives:

Primary objectives:

* To determine if neoadjuvant chemotherapy with or without panitumumab followed by deferred surgery and completion of chemotherapy postoperatively can reduce the 2-year recurrence as compared to surgery and postoperative chemotherapy with or without panitumumab.
* To determine if, in patients with RAS-wt tumours, adding panitumumab to neoadjuvant therapy increases anti-tumour activity as measured by tumour shrinkage.

Secondary

* To assess the accuracy of pre-treatment CT scan staging.
* To assess the tolerability of the neoadjuvant therapies.
* To assess the nature and frequency of surgical complications.
* To measure the impact of the treatments on quality of life and on resource usage.
* To assess whether adding panitumumab to neoadjuvant CT reduces 2-year recurrence
* To assess the prognostic and predictive value of tumour biomarkers
* To assess the influence of resectional quality on outcome

OUTLINE: This is a multicenter study. Patients are stratified according to age (< 50 year vs 50-59 years vs 60-69 years vs ≥ 70 years), radiological T-stage (T3 vs T4), radiological nodal status (Nx vs N0 vs N1 vs N2), site of primary tumor, proposed chemotherapy (OxMdG vs OxCap), and defunctioning colostomy (yes vs no). Planned chemo duration 12 or 24 weeks.

Patients receive 1 of the 2 following treatment regimens:

* OxMdG: Patients receive oxaliplatin IV and folinic acid IV over 2 hours followed by fluorouracil IV continuously over 46 hours on day 1 for 1 course.
* OxCap: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-15 for 1 course.

Patients are randomized to 1 of 2 treatment arms.

* Neoadjuvant therapy:

  * Arm I: Patients receive 1 of the following chemotherapy regimens:

    * OxMdG: Patients receive oxaliplatin IV over 2 hours and fluorouracil IV continuously over 46 hours on day 1. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
    * OxCap: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-15. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive the following regimen:

    * OxMdG + panitumumab: Patients receive panitumumab IV over 60 minutes on day 1 followed by oxaliplatin IV over 2 hours and fluorouracil IV continuously over 46 hours on day 1. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Approximately 52 days after beginning chemotherapy, patients in both arms proceed to surgery.

* Surgery: Patients in both arms undergo surgical resection of the primary tumour.
* Adjuvant therapy: Beginning 4-8 weeks after completion of surgery, patients receive adjuvant treatment on the same arm for which they received neoadjuvant therapy.

  * Patients receive either nine 2-week courses of OxMdG therapy or six 3-week courses of OxCap therapy.

Tumour tissue is collected during surgery and blood samples are collected periodically for biomarker studies. Samples are analyzed for the detection of KRAS and NRAS mutations; the detection of EGFR expression and/or functional genetic polymorphisms of the EGFR gene via PCR; the detection of copy number EGFR gene amplification via fluorescence in situ hybridization (FISH); the detection of EGFR activation via immunohistochemistry (IHC); the detection of EGFR by downstream parameters via western blotting and/or gene expression microarray techniques; for proteomics; and for epigenetics.

Patients complete quality of life questionnaires prior to surgery, before first course of postoperative chemotherapy, and at 1 year following randomization.

After completion of study treatment, patients are followed every 6 months for 3 years and then annually thereafter.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically proven adenocarcinoma of the colon or high grade dysplasia on histology plus unequivocal radiological evidence of invasive cancer.
* A candidate for adjuvant oxaliplatin/ fluoropyrimidine chemotherapy based on:

  * Either radiological high risk (rT4 or rT3 tumour with extramural extension ≥ 5mm)
  * Or radiological intermediate risk (rT3 tumour with <5mm extramural extension) and younger age/good general health
* Patients presenting with acute colonic obstruction may enter the trial only after obstruction is relieved by a successful defunctioning stoma, and when recovered to a fitness level consistent with the other eligibility criteria
* Adequate full blood count: WBC >3.0 x109/l; Plts >100 x109/l. Anaemia (Hb < 10.0 g/dl) is not an exclusion, but should be corrected by transfusion prior to surgery and chemotherapy. If Hb remains low despite transfusions, surgery and chemotherapy can be given at the decision of the surgical and oncology teams.
* Adequate renal biochemistry: GFR >50 ml/min calculated by the Wright or Cockroft formula or EDTA clearance >70 ml/min
* Adequate hepatobiliary function: bilirubin < 25 μmol/l (Patients with Gilbert's syndrome who have raised bilirubin but otherwise normal liver function tests are eligible for the study.)
* Aged 18 or over
* WHO performance status of 0, 1 or 2
* If female and of childbearing potential, must:

  * Have a negative pregnancy test ≤72hours prior to initiating study treatment
  * Agree to avoid pregnancy during and for 6 months after study treatment
* If male with a partner of childbearing potential, must:

  - Agree to use adequate, medically approved, contraceptive precautions during and for 90 days after the last dose of study treatment
* Patient able and willing to provide written informed consent for the study

EXCLUSION CRITERIA

* Any patient for whom radiotherapy is advised by the MDT
* Strong evidence of distant metastases or peritoneal nodules (M1)
* Peritonitis (secondary to perforated tumour)
* Colonic obstruction that has not been defunctioned
* Serious medical comorbidity, eg uncontrolled inflammatory bowel disease, uncontrolled angina or recent (<6 months) MI
* Another serious medical condition judged to compromise ability to tolerate neoadjuvant therapy and/or surgery
* Any other malignant disease within the preceding 5 years with the exception of non-melanomatous skin cancer, carcinoma in situ and early stage disease with a recurrence risk <5%

ADDITIONAL EXCLUSION CRITERIA FOR PANITUMUMAB RANDOMISATION

* RAS-mutant or unknown RAS status tumours
* Allocated post-operative chemotherapy
* History of interstitial pneumonitis or pulmonary fibrosis
* History of severe or life-threatening hypersensitivity reactions
* Serum magnesium levels within the normal range at trial entry (which can include intravenous correction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2008-05-15 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from recurrence or persistent disease (including failure of macroscopic disease clearance at primary surgery) within the first two years following randomization | 2 year post randomization
Pathological down-staging as measured by depth of extramural spread among patients allocated to preoperative chemotherapy with or without panitumumab | Time of surgery

SECONDARY OUTCOMES:
Death from colon cancer | 2 years
Overall survival | 2 years
Freedom from recurrence or persistent disease at 2 years (panitumumab comparison) | 2 years
Pathological assessment of downstaging (involvement of lymph nodes, serosa, and resection margin) and quality of resection specimen | at surgery
Quality of resection specimen and distance to high-tie | post surgery
Radiological assessment of response to neoadjuvant treatment | prior to surgery
Quality of life by EORTC QLQ C-30 and EuroQol EQ-5D | before surgery, before 1st post-op chemo, 1 year post randomization
Lenght of hospital stay | post surgery
Surgical morbidity/mortality | 30 days post surgery
Chemotherapy toxicity | during chemotherapy administration
Adverse events | throughout the trial, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dion Morton, MD, Principal Investigator — University of Birmingham
Locations (10):
- United Kingdom (10):
  - Birmingham Clinical Trials Unit, Birmingham, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Clatterbridge Centre for Oncology, Metropolitan Borough of Wirral, England
  - Derriford Hospital, Plymouth, England
  - Southport and Formby District General Hospital, Southport, England
  - Sandwell General Hospital, West Bromwich, England

REFERENCES:
- [Derived] FOxTROT Collaborating Group. Risk of Bowel Obstruction in Patients Undergoing Neoadjuvant Chemotherapy for High-risk Colon Cancer: A Nested Case-control-matched Analysis of an International, Multicenter, Randomized Controlled Trial (FOxTROT). Ann Surg. 2024 Aug 1;280(2):283-293. doi: 10.1097/SLA.0000000000006145. Epub 2023 Nov 10. PMID 37947140
- [Derived] Morton D, Seymour M, Magill L, Handley K, Glasbey J, Glimelius B, Palmer A, Seligmann J, Laurberg S, Murakami K, West N, Quirke P, Gray R; FOxTROT Collaborative Group. Preoperative Chemotherapy for Operable Colon Cancer: Mature Results of an International Randomized Controlled Trial. J Clin Oncol. 2023 Mar 10;41(8):1541-1552. doi: 10.1200/JCO.22.00046. Epub 2023 Jan 19. PMID 36657089
- [Derived] van den Berg I, Smid M, Coebergh van den Braak RRJ, van de Wiel MA, van Deurzen CHM, de Weerd V, Martens JWM, IJzermans JNM, Wilting SM. A panel of DNA methylation markers for the classification of consensus molecular subtypes 2 and 3 in patients with colorectal cancer. Mol Oncol. 2021 Dec;15(12):3348-3362. doi: 10.1002/1878-0261.13098. Epub 2021 Sep 30. PMID 34510716
- See also: Feasibility of preoperative chemotherapy for locally advanced, operable colon cancer: the pilot phase of a randomised controlled trial. Lancet Oncol. 2012 Nov;13(11):1152-60. doi: 10.1016/S1470-2045(12)70348-0. Epub 2012 Sep 25. — http://www.ncbi.nlm.nih.gov/pubmed/23017669
- See also: FOxTROT website — http://www.birmingham.ac.uk/FOxTROT